CLINICAL TRIAL: NCT06796660
Title: Exploring the Impact of Nephropathy Formula No. 1 on T-Cell Immune Balance in Chronic Kidney Disease Patients Via the IL-6/STAT3 Signaling Pathway
Brief Title: Exploring the Impact of Nephropathy Formula No. 1 on Chronic Kidney Disease Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Liu Zhanghong (Other)
Responsible Party: Sponsor-Investigator, Liu Zhanghong, Deputy Chief physician of Traditional Chinese Medicine, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZL081
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Integrated Basic Treatment for Chronic Kidney Disease (CKD) Can Utilize the Following ：α-Keto acid tablets (2.6 g tid) ；Antihypertensive drugs such as amlodipine tablets (5 mg qd), nifedipine tablets (30 mg qd), or losartan tablets (100 mg qd)；Medications such as repaglinide tablets (1.0 mg qd) or gliclazide modified-release tablets (30 mg qd) ；Medications such as atorvastatin calcium tablets (20 mg qd) or fenofibrate capsules (0.2 g qd)； Recombinant human erythropoietin (10000 u qw)； Composition and Preparation of Nephropathy Formula No. 1 includes: Bupleurum , Paeonia lactiflora Pall. , Scutellaria baicalensis Georgi , Pinellia ternata (Thunb.) Breit. , Smilax glabra Roxb. , Oldenlandia diffusa (Willd.) Roxb. , Rhus chinensis Mill. , and Poria cocos (Schw.) Wolf . The decoction is concentrated to 300 ml, with one dose per day, taken in two divided doses.The treatment period for the above regimen is 12 weeks.
  Interventions: Drug: Nephropathy Formula No. 1; Drug: integrated basic treatment for chronic kidney disease
- Control Group (Active Comparator): The control group will receive integrated basic treatment for chronic kidney disease, including: ① Nutritional diet with low salt, low fat, and low high-quality protein, with a protein intake of 0.6-0.8g/(kg·d), of which 50% comes from high-quality protein, and essential amino acids or α-keto acid preparations of 0.1-0.2g/(kg·d) are supplemented. ② Blood pressure control. ③ Blood sugar control. ④ Lipid control. ⑤ Anemia treatment. ⑥ Regulation of water, electrolyte, and acid-base metabolic balance.
  Interventions: Drug: integrated basic treatment for chronic kidney disease

INTERVENTIONS:
Drug: Nephropathy Formula No. 1 — On the basis of integrated treatment for chronic kidney disease (the specific plan is the same as the control group), Nephropathy Formula No. 1 is given orally. The composition and decoction method of the formula are as follows: Bupleurum, Paeonia lactiflora Pall. , Scutellaria baicalensis Georgi , Pinellia ternata (Thunb.) Breit. , Smilax glabra Roxb. , Oldenlandia diffusa (Willd.) Roxb. , Tussilago farfara L. , Poria cocos (Schw.) Wolf , decocted into 300ml, one dose per day, taken warm in two divided doses for 12 weeks.
  Other Names: Administration group
  Arms: Treatment group
Drug: integrated basic treatment for chronic kidney disease — The integrated basic treatment for CKD includes the following:
  Dietary Nutrition: α-Keto acid tablets (2.6 g tid) may be used. Blood Pressure Control: Antihypertensive drugs such as amlodipine tablets (5 mg qd), nifedipine tablets (30 mg qd), or losartan tablets (100 mg qd) can be selected. β-blockers or α-blockers may be used in combination if necessary.
  Blood Sugar Control: Medications such as repaglinide tablets (1.0 mg qd) or gliclazide modified-release tablets (30 mg qd) can be used.
  Lipid Control: Medications such as atorvastatin calcium tablets (20 mg qd) or fenofibrate capsules (0.2 g qd) can be used.
  Anemia Treatment: Recombinant human erythropoietin (10000 u qw) can be administered via subcutaneous injection.
  Regulation of Water, Electrolyte, and Acid-Base Metabolic Balance.
  Other Names: control group

SUMMARY:
This study is a prospective randomized controlled trial, enrolling 70 patients with CKD stages 2-4, randomly divided into a control group and a treatment group, with 35 cases in each group. The study subjects are sourced from three centers. The control group receives integrated basic treatment for chronic kidney disease, including dietary nutrition adjustment, blood pressure control, blood sugar control, lipid control, anemia treatment, and regulation of water, electrolyte, and acid-base metabolic balance. The treatment group, in addition to the basic treatment, is administered Nephropathy Formula No. 1 orally, with a treatment course of 12 weeks and a follow-up period of 2 weeks. The outcome measures are the changes in biochemical indicators, inflammatory factors, T cell subsets, STAT3 mRNA expression, and TCM syndrome scores after 12 weeks of treatment, to assess therapeutic efficacy. This study proposes the experimental hypothesis that Nephropathy Formula No. 1 can effectively improve the T cell immune balance in CKD patients by modulating the IL-6/STAT3 signaling pathway, thereby inhibiting the occurrence and development of renal fibrosis and improving the prognosis of CKD to a certain extent. Specifically, Nephropathy Formula No. 1 may function through the following mechanisms: (1) downregulating IL-6 mRNA expression, reducing IL-6 secretion, and thereby inhibiting the activation of the STAT3 signaling pathway; (2) regulating the balance of Th17/Treg cell subsets, promoting the differentiation of Th17 cells into Treg cells, enhancing the anti-inflammatory and immunosuppressive effects of Treg cells, and alleviating renal inflammatory responses and fibrosis. Through in-depth exploration of this study, it is expected to provide new ideas and methods for the clinical treatment of CKD, with significant scientific and clinical implications.

DETAILED DESCRIPTION:
Sample Size Estimation Sample size estimation is based on the results of a pilot study. A total of 60 patients are required for enrollment. Considering a dropout rate of 10%-15%, each group will need 35 cases, with a total of 70 cases for both groups.

Patient Recruitment Patients will be recruited by researchers during outpatient or inpatient visits. After screening according to the inclusion and exclusion criteria, eligible patients will be enrolled in the study following the signing of the informed consent form.

Adverse Events and Serious Adverse Events Management Severity: Physicians can use the following definitions to judge the severity of all adverse events and serious adverse events, which will serve as endpoints/data cutoff points for the study.

Mild: Adverse events are transient and easily tolerated by the patient. Moderate: Adverse events cause discomfort to the subject and interfere with their normal activities.

Severe: Adverse events significantly impact the subject's daily activities and may result in functional loss or be life-threatening.

Management of Adverse Events: In the clinical trial, if any adverse event occurs, regardless of its causal relationship with the investigational drug or the treatment method used, the researcher must take necessary measures for treatment and rescue. For adverse events that occur during the trial, the type, severity, onset time, duration, management measures, and course of action should be recorded in the inpatient medical record and the case report form. A comprehensive analysis should be conducted to determine whether the event is related to the trial. After an adverse event occurs, the researcher may decide whether the subject should discontinue the clinical trial based on the condition. For cases terminated due to serious adverse events, follow-up and recording of their outcomes should be conducted.

Recording and Reporting of Serious Adverse Events: If a serious adverse event occurs during the trial, regardless of its relationship to the trial, immediate emergency measures should be taken, and the principal investigator and the ethics committee should be notified by phone within 24 hours. Subsequently, a serious adverse event report form should be completed and promptly submitted to the aforementioned departments.

Monitoring and Recording of Adverse Events This includes any symptoms, signs, and laboratory abnormalities that occur from the time of signing the informed consent form to the end of the last visit. The occurrence of adverse events should be specifically described, including the time of occurrence, severity, duration, measures taken, and outcome. All adverse events should be recorded in the designated case report form for adverse events.

Data Management Researchers are required to fill in the collected data into the case report form according to the study protocol and use EXCEL software for data collection or recording. Data management will be handled by a designated person to ensure the authenticity, completeness, and accuracy of the clinical trial data. At the end of the study, researchers will submit all the case report forms of the enrolled patients to the data management center. These case report forms should be complete and signed. Consistency of data collected from various research centers will be checked, and queries will be issued for any inconsistencies, which the researchers will need to clarify. Missing data will be preserved but not included in the statistical analysis.

Data Description Quantitative data will be described using mean ± standard deviation (SD), median, maximum, minimum, and quartiles. Categorical data will be represented as percentages (%).

Data Statistics All statistical tests, unless otherwise specified, will use a two-sided test. A P-value of less than 0.05 will be considered statistically significant. Comparisons of general conditions among groups will be analyzed using appropriate methods based on data type and distribution. For example, comparisons of quantitative indicators between groups will use one-way analysis of variance (ANOVA) (for homoscedasticity and normal distribution) or the Kruskal-Wallis rank-sum test (for non-normal distribution); categorical indicators will use the chi-square test or Fisher's exact test (if the chi-square test is not applicable), and ordinal indicators will use the Kruskal-Wallis rank-sum test or the Cochran-Mantel-Haenszel (CMH) test. A P-value of less than 0.05 will be considered statistically significant.

Statistical Analysis Plan This will be completed by professional statisticians. After all data entry and review are completed, statisticians should promptly conduct the statistical analysis and produce a written statistical analysis report.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old (inclusive);
2. No gender restriction;
3. Patients diagnosed with CKD stages 2-4 according to the above diagnostic criteria by a specialist physician;
4. TCM syndrome differentiation is consistent;
5. Able to cooperate with the study treatment and follow-up, and has good compliance;
6. Agree and sign the medical informed consent form.

Exclusion Criteria:

1. Patients undergoing hemodialysis or peritoneal dialysis;
2. Patients with severe primary diseases of the cardiovascular, hematological, digestive, nervous, respiratory, endocrine systems, malignant tumors, etc.;
3. Patients in the active phase of autoimmune system diseases;
4. Patients with chronic infectious diseases such as active viral hepatitis, HIV, or active tuberculosis;
5. Patients with recent acute infections, and non-infectious complications such as hypertension and anemia that have not been effectively controlled;
6. Patients who have taken traditional Chinese medicine related to nephropathy treatment within the past month;
7. Patients who have undergone surgery, trauma, major bleeding, or blood transfusion within the past three months, or have severe clinical infections, electrolyte disturbances, and acid-base imbalances that have not been effectively controlled;
8. Pregnant or breastfeeding women;
9. Patients with mental disorders or poor compliance who cannot cooperate;
10. Patients who have participated in other drug tests within the past three months or have not completed the effective drug washout period. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the ratio of Th17 to Treg cells in T cell subsets | 12 weeks
  The ratio of Th17 to Treg cells in peripheral blood will be measured using flow cytometry. The Th17/Treg ratio will be compared before and after treatment to determine the experimental outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanghong Z Liu, Master, Principal Investigator — The Third Afffliated Hospital of Zhejiang Chinese Medical University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Wenzhou TCM Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Wenzhou TCM Hospital of Zhejiang Chinese Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No